CLINICAL TRIAL: NCT01422915
Title: Sorbent Therapy of the Cutaneous Porphyrias
Acronym: EPP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Peter Tishler, physician, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010P002253
Record Dates: First submitted 2011-08-23; First posted 2011-08-25 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-03

CONDITIONS: Erythropoietic Protoporphyria
Keywords: Sorbent; Resin; EPP; Cutaneous porphyria; Adult; over age 21; without intercurrent illness; not pregnant; willing to participate
MeSH Terms: conditions — Protoporphyria, Erythropoietic | interventions — Colestipol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- colestipol treatment (Experimental): 2 grams morning and bedtime for 180 days
  Interventions: Drug: Colestipol

INTERVENTIONS:
Drug: Colestipol — 2 grams morning and bedtime for 90 days.

SUMMARY:
The investigators demonstrated that cholestyramine is an effective binding agent in vitro for porphyrins. A few isolated case reports of treatment of individuals with a cutaneous porphyria suggest that cholestyramine and colestipol effectively remove porphyrins. Hypothesis: orally administered colestipol will effectively reduce sun sensitivity and lower erythrocyte porphyrin concentrations in subjects with erythropoietic protoporphyria (EPP).

DETAILED DESCRIPTION:
Four adults with proven EPP volunteered as subjects for this study. First period: Subjects received 1 gm colestipol twice daily for ~45 days, then 2 gm twice daily for ~45 days. Labs included CBC; liver chemistries including cholesterol; serum iron, TIBC and ferritin; erythrocyte and plasma protoporphyrin concentrations; and completion of sun exposure questionnaire focused on cutaneous manifestations every 2-4 weeks. Second period: Subjects received colestipol tablets, 2 grams twice daily, completing the sun exposure questionnaire and protoporphyrin determinations ~monthly for 5-6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult over age 21
* healthy

Exclusion Criteria:

* Intercurrent illness
* pregnancy

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2011-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates: February and March 2011.Location types: suburbs of Massachusetts (3 subjects) and in New Jersey (1).
Pre-assignment Details: All 4 subjects were enrolled in the study. Initially, baseline blood protoporphyrin concentrations and answers to sun sensitivity questionnaire were obtained.
Groups:
- Colestipol Treatment: Colestipol 2 grams twice daily for 5-6 months. Completion of sun sensitivity questionnaire and blood protoporphyrin concentrations. were obtained monthly.
Period: Overall Study
Arm/Group | Colestipol Treatment
Started | 4 (1 subject with abnormal liver chemistries removed during the first period.)
Completed | 3
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Colestipol Therapy of Protoporphyria: 4 subjects were assigned, all between 18-65 years of age.
Arm/Group | Colestipol Therapy of Protoporphyria
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (15)
Age, Customized [Number; unit: participants] — For baseline in Period 1 and Period 2: ~monthly completion of sun sensitivity questionnaire; donate whole blood for RBC and plasma protoporphyrin
  participants
    <=18 years | 0
    Between 18 and 65 years | 4
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Photosensitivity, Assessed by Measuring the Number of Minutes of Sun Tolerance
Description: Minutes of sun tolerance
Time Frame: At 60 days of treatment
Population: All of the original 4 subjects had bona fide erythropoietic protoporphyria (EPP). One subject was removed during Perdiod 1. The data from the same 3 subjects who completed periods 1 and 2 were analyzed for the study results. Data collected was not tractable for statistical analysis given the range of results
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Colestipol Treatment: 1. gram morning and bedtime for 90 days; then
  2. grams morning and bedtime for 90 days. Sun sensitivity questionnaires and blood protoporphyrin concns. were determined monthly.
Arm/Group | Colestipol Treatment
Number analyzed (Participants) | 3
minutes | 65.8 (58.8)

2. Primary Outcome: Protoporphyrin Concentration in Blood
Description: 1. erythrocyte protoporphyrin concentration, ug/dl
  2. plasma protoporphyrin concentration, ug/dl
Time Frame: Samples collected while on treatment (range 93-208 treatment days)
Measure: Mean (Standard Deviation); unit: ug/dl
Groups:
- Colestipol Treatment: Sun sensitivity and protoporphyrin levels
Arm/Group | Colestipol Treatment
Number analyzed (Participants) | 3
ug/dl
  Erythrocyte Protoporphyrin | 1712 (455)
  Plasma Protoporphyrin | 5.8 (8.3)

ADVERSE EVENTS:
Groups:
- 1st Period - Colestipol Optimal Dosage: 1. gram morning and bedtime for 90 days; then
  2. grams morning and bedtime for 90 days. Sun sensitivity questionnaires and blood protoporphyrin concentrations were determined monthly.
Arm/Group | 1st Period - Colestipol Optimal Dosage
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1st Period - Colestipol Optimal Dosage (N=4)
Abnormal liver enzymes (Hepatobiliary disorders) | 1 (1) — Abnormal liver enzymes on one occasion.

LIMITATIONS AND CAVEATS:
1 subject was removed during Period 1 because of abnormal liver chemistries.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No